CLINICAL TRIAL: NCT03542539
Title: The Role of Dermoscopy in Diagnosis of Pigmentary Skin Lesions
Brief Title: Dermoscopy in Diagnosis of Pigmentary Skin Lesions
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Sobeith, principal investigator, Assiut University
Other Study IDs: RODIPSL
Record Dates: First submitted 2018-03-26; First posted 2018-05-31 (Actual); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Pigmentary Skin Lesions; Dermoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Dermoscopy is a non-invasive method that allows evaluation of colors and microstructures of the epidermis, the dermoepidermal junction, and the papillary dermis not visible to the naked eye. These structures are specifically correlated to histologic features. The identification of specific diagnostic patterns related to the distribution of colors and dermoscopy structures can better suggest a malignant or benign pigmented skin lesion. The use of this technique provides a valuable aid in diagnosing pigmented skin lesions

DETAILED DESCRIPTION:
Skin color affected by many agents as it is determined by several chromophores such as melanin, hemoglobin and carotenoids. Among these, melanin is the main one responsible for different skin colors.

Melanin is produced by special skin cells called melanocytes and packed in organelles called melanosomes. Sometimes, human skin may present a non-uniform melanin distribution in two different ways, leading to pigmentary disorders.

In the first, melanin concentration increases to levels above normal resulting in hypermelanosis. In the second, the melanin concentration decreases to levels below normal, resulting in hypomelanosis.melanogenesis is acomplex process when disturbed ,it results into various pigmentary disorders either hypo or hyper pigmentation.

These disorders may be congenital or acquired, permenant or temporary, systemic or region restricted).

Pigmentary disorders are include alarge number of heterogenous conditions that are usually characterized by altered melanocyte density, melanin concentration, or both, and result in altered pigmentation of the skin. Some of these disorders are extremely common such as (melisma and vitiligo), whereas others are rare

Differential Diagnosis of Hyper and Hypopigmentation:

Hyperpigmentation Hypopigmentation Postinflammatory hyperpigmentation (acne, psoriasis, atopic and contact dermatitis, lichen planus, trauma, drugs, and fixed-drug eruptions) Melasma Solar lentigines Ephelides (freckles) Café-au-lait macules Nevi Melanoma and precursors Acquired (common) Vitiligo Pityriasis alba Tinea versicolor Postinflammatory hypopigmentation Congenital (uncommon) Albinism Piebaldism Tuberous sclerosis Hypomelanosis of Ito

Several studies have shown that dermoscopy may come in very handy for assisting the noninvasive diagnosis of various general dermatological disorders, including scalp/hair diseases (trichoscopy) , nail/nailfold abnormalities (onychoscopy) , cutaneous infections/infestations (entomodermoscopy) and inflammatory dermatoses (inflammoscopy) .

Dermoscopy is a non-invasive method that allows evaluation of colors and microstructures of the epidermis, the dermoepidermal junction, and the papillary dermis not visible to the naked eye. These structures are specifically correlated to histologic features. The identification of specific diagnostic patterns related to the distribution of colors and dermoscopy structures can better suggest a malignant or benign pigmented skin lesion. The use of this technique provides a valuable aid in diagnosing pigmented skin lesions, This traditionally consists of a magnifier , a non-polarised light source, a transparent plate and a liquid medium between the instrument and the skin .

The increasing use of dermoscopy in general dermatology can be partially explained by commercially available new generations of handheld dermoscopes, which are small enough to be easily placed in every dermatologist's pocket . It is a safe and rapid diagnostic tool that assists in clinical examination and management decision in dermatology

ELIGIBILITY:
Inclusion Criteria:

* all patients attending assuit university hospital clinics complaining of pigmentary skin lesions

Exclusion Criteria:

* no exclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: all patients attending assiut university hospital clinics complaining of pigmentary skin lesions
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients with pigmentary lesions | 24 hours
  use of dermoscope for diagnosis